CLINICAL TRIAL: NCT01227902
Title: An Open-Label, Flexible-Dose Study of Retigabine Immediate Release (IR) as Adjunctive Therapy to Specified Monotherapy Antiepileptic Treatments in Adults With Partial -Onset Seizures
Brief Title: Study of Retigabine Immediate Release as Adjunctive Therapy to Specified Monotherapy Antiepileptic Treatments in Adults With Partial-Onset Seizures
Acronym: IR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 113905
Record Dates: First submitted 2010-07-16; First posted 2010-10-25 (Estimated); Results first posted 2013-11-11 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Epilepsy
Keywords: Seizures; retigabine IR; GW582892; Epilepsy; Open label, flexible dose; Partial-onset seizures
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Retigabine IR (Experimental): Open Label flexible dose between 300 mg/day (minimum) and 1200 mg/day (maximum).
  Interventions: Drug: Retigabine IR

INTERVENTIONS:
Drug: Retigabine IR — Flexible dose between 300 mg/day (minimum) and 1200 mg/day (maximum).

SUMMARY:
The purpose of this Phase III study is to evaluate the efficacy, safety and tolerability and health outcomes of retigabine Immediate Release (IR) as adjunctive therapy to each of the following monotherapy Antiepileptic Drug (AED) treatments: carbamazepine/oxcarbazepine, lamotrigine, levetiracetam, or valproic acid in adult subjects with partial-onset seizures (POS) using a flexible dosing regimen.

DETAILED DESCRIPTION:
This is an open-label, multi-centre, flexible dose study of retigabine immediate release (IR). The study will enroll male and female outpatients (≥ 18 years of age) with partial-onset seizures (POS) who are inadequately controlled on their current monotherapy Antiepileptic Drug (AED). Following a Screening Period of up to 2 weeks, subjects will enter an 8-week Baseline Phase to determine baseline seizure frequency. At the end of the Baseline Phase, subjects who meet or exceed the minimum seizure frequency of 4 partial seizures per 56 days, will enter the Treatment Period (4 weeks Titration, 16 weeks Flexible Dose Evaluation Phase). All subjects will receive retigabine IR starting at 150 mg/day and will be titrated to 600 mg/day by Week 4. From Week 5 onwards, subjects' doses will be maintained between 300 to 1200 mg/day using a flexible dosing regimen to optimise response and tolerability. The maximum duration of the study is approximately 33 weeks (inclusive of a 3 week Taper/Follow-up Phase).

ELIGIBILITY:
Inclusion Criteria:

* Is 18 years of age (men or women)
* Has a confident diagnosis of epilepsy with partial-onset seizures i.e., simple or complex partial seizures with or without secondary generalization (International League Against Epilepsy (ILAE) classification; 1981) for more than 24 weeks prior to the start of Baseline phase.
* Has experienced at least 4 partial-onset seizures (i.e., simple or complex partial seizures with or without secondary generalization) during an 8-week (i.e., 56 days) prospective Baseline Phase with at least one partial seizure occurring during each 4 week (i.e., 28-day) period.
* Receiving a stable dose of one of the following AEDs: carbamazepine/oxcarbazepine, lamotrigine, levetiracetam or valproic acid. The AED dose must be stable 4 weeks prior to start of collection of baseline seizure data (retrospective or prospective) and during the Baseline period.
* Is able and willing to maintain an accurate and complete daily written seizure calendar and functional status diary or has a caregiver who is able and willing to do so for the entire duration of the study.
* Is able to comply with dosing of study drug, background AED and all study procedures.
* Has given written informed consent, or has a legally authorized representative who has given written informed consent, prior to the performance of any study assessments.
* A female subject is eligible to enter and participate in the study if she is either of non-childbearing potential or child-bearing potential but has a negative pregnancy test at Screening and agrees to satisfy one of the contraception methods as listed in the protocol, and is not pregnant or lactating or planning to become pregnant during the study.
* French subjects only: In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.

Exclusion Criteria:

* Has a history of generalised epilepsy (e.g. Lennox-Gastaut, Juvenile Myoclonic etc.)
* Has had status epilepticus (other than simple partial status epilepticus) within the 24 weeks prior to Baseline Visit.
* Has participated in a previous retigabine study (subjects with documented evidence of having received placebo will be eligible).
* Is currently or has been abusing substance(s) or other medications in the 12 months prior to Baseline visit.
* Has taken an investigational drug, or used an investigational device, within the previous 30 days prior to screening or plans to take an investigational drug anytime during the study.
* Is currently following or planning to follow the ketogenic diet.
* Has been treated with vigabatrin within the past 6 months prior to collection of baseline seizure data.
* Is planning surgery or implantation of a Vagus Nerve Stimulator (VNS) to control seizures during the study.
* Is suffering from acute or progressive neurological disease, severe psychiatric disease, or severe mental abnormalities that are likely to interfere with the objectives of the study.
* Has any medical condition that, in the investigator's judgment, is considered to be clinically significant and could potentially affect subject safety or study outcome.
* Has a QTc ≥450 millisecond (msec) or greater than or equal to 480 msec for subjects with Bundle Branch Block at the time of screening.
* Has active suicidal plan/intent or has had active suicidal thoughts in the past 6 months. Has history of suicide attempt in the last 2 years or more than 1 lifetime suicide attempt.
* French Subjects: the French subject has participated in any study using an investigational drug during the previous 30 days or 5 half-lives (whichever is longer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2010-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (62):
- Belgium (3):
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Liège
- Bulgaria (3):
  - GSK Investigational Site, Pleven
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Sofia
- Denmark (3):
  - GSK Investigational Site, Dianalund
  - GSK Investigational Site, Glostrup Municipality
  - GSK Investigational Site, Koebenhavn Oe
- France (6):
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Limoges
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Nancy
  - GSK Investigational Site, Rennes
  - GSK Investigational Site, Strasbourg
- Germany (8):
  - GSK Investigational Site, Kehl-Kork, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Tübingen, Baden-Wurttemberg
  - GSK Investigational Site, Marburg, Hesse
  - GSK Investigational Site, Bielefeld, North Rhine-Westphalia
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Kiel, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin
- Italy (9):
  - GSK Investigational Site, Foggia, Apulia
  - GSK Investigational Site, Reggio Calabria, Calabria
  - GSK Investigational Site, Bologna, Emilia-Romagna
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Palermo, Sicily
  - GSK Investigational Site, Torrette Di Ancona, The Marches
  - GSK Investigational Site, Pisa, Tuscany
  - GSK Investigational Site, Siena, Tuscany
- Netherlands (4):
  - GSK Investigational Site, Breda
  - GSK Investigational Site, Heemstede
  - GSK Investigational Site, Heeze
  - GSK Investigational Site, The Hague
- Poland (4):
  - GSK Investigational Site, Iława
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Warsaw
- Russia (7):
  - GSK Investigational Site, Belgorod
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Krasnodar
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Samara
  - GSK Investigational Site, Smolensk
- Spain (4):
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Vigo
- Thailand (3):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Khon Kaen
  - GSK Investigational Site, Songkhla
- Ukraine (8):
  - GSK Investigational Site, Dnipro
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Luhansk
  - GSK Investigational Site, Lviv
  - GSK Investigational Site, Odesa
  - GSK Investigational Site, Oleksandrivka Village, Odesa
  - GSK Investigational Site, Poltava

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study 113905 was an open-label, multi-center, multi-country study of retigabine using a flexible dosing regimen in adult participants (>=18 years old) with partial-onset seizures. Eligible participants must have been taking one of the following antiepileptic drug treatments: carbamazepine/oxcarbazepine, lamotrigine, levetiracetam, or valproic acid.
Pre-assignment Details: Eligible participants were required to have had at least 4 partial seizures during the 8-week Baseline Phase and must have been receiving a stable dose of one of the prespecified monotherapy antiepileptic drug treatments.
Groups:
- RTG Flexible Dose Plus C/O: Along with concurrent carbamazepine/oxcarbazepine (C/O), participants initiated treatment with retigabine (RTG) immediate release (IR) at 150 milligrams per day (mg/day) (50 mg thrice a day [TID]) and titrated to 600 mg/day (200 mg/day TID) over a 4-week Titration Phase. This was followed by a 16-week Flexible Dose Evaluation Phase, during which the dose could be increased or decreased on a weekly basis between 50 and 150 mg/day, depending on efficacy and tolerability, with the total dose staying between 300 and 1200 mg/day. Participants who were unable to tolerate a minimum dose of 300 mg/day were discontinued from the study.
- RTG Flexible Dose Plus Lamotrigine: Along with concurrent lamotrigine, participants initiated treatment with RTG IR at 150 mg/day (50 mg TID) and titrated to 600 mg/day (200 mg/day TID) over a 4-week Titration Phase. This was followed by a 16-week Flexible Dose Evaluation Phase, during which the dose could be increased or decreased on a weekly basis between 50 and 150 mg/day, depending on efficacy and tolerability, with the total dose staying between 300 and 1200 mg/day. Participants who were unable to tolerate a minimum dose of 300 mg/day were discontinued from the study.
- RTG Flexible Dose Plus Levetiracetam: Along with concurrent leveteracetam, participants initiated treatment with RTG IR at 150 mg/day (50 mg TID) and titrated to 600 mg/day (200 mg/day TID) over a 4-week Titration Phase. This was followed by a 16-week Flexible Dose Evaluation Phase, during which the dose could be increased or decreased on a weekly basis between 50 and 150 mg/day, depending on efficacy and tolerability, with the total dose staying between 300 and 1200 mg/day. Participants who were unable to tolerate a minimum dose of 300 mg/day were discontinued from the study.
- RTG Flexible Dose Plus Valproic Acid: Along with concurrent valproic acid, participants initiated treatment with RTG IR at 150 mg/day (50 mg TID) and titrated to 600 mg/day (200 mg/day TID) over a 4-week Titration Phase. This was followed by a 16-week Flexible Dose Evaluation Phase, during which the dose could be increased or decreased on a weekly basis between 50 and 150 mg/day, depending on efficacy and tolerability, with the total dose staying between 300 and 1200 mg/day. Participants who were unable to tolerate a minimum dose of 300 mg/day were discontinued from the study.
Period: Overall Study
Arm/Group | RTG Flexible Dose Plus C/O | RTG Flexible Dose Plus Lamotrigine | RTG Flexible Dose Plus Levetiracetam | RTG Flexible Dose Plus Valproic Acid
Started | 56 | 51 | 44 | 52
Completed | 38 | 38 | 25 | 42
Not Completed | 18 | 13 | 19 | 10
Not completed — Adverse Event | 12 | 8 | 11 | 4
Not completed — Lack of Efficacy | 1 | 2 | 2 | 1
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 2
Not completed — Physician Decision | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 4 | 2 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RTG Flexible Dose Plus C/O | RTG Flexible Dose Plus Lamotrigine | RTG Flexible Dose Plus Levetiracetam | RTG Flexible Dose Plus Valproic Acid | Total
Number analyzed (Participants) | 56 | 51 | 44 | 52 | 203
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline data were collected in members of the Safety Population, comprised of those participants who took at least one dose of RTG.
  Years | 40.6 (14.99) | 38.2 (11.91) | 37.0 (14.94) | 40.3 (14.05) | 39.1 (14.00)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline data were collected in members of the Safety Population, comprised of those participants who took at least one dose of RTG.
  Participants
    Female | 33 | 26 | 25 | 26 | 110
    Male | 23 | 25 | 19 | 26 | 93
Race/Ethnicity, Customized [Number; unit: participants] — Baseline data were collected in members of the Safety Population, comprised of those participants who took at least one dose of RTG.
  participants
    Asian - Central/South Asian Heritage | 1 | 1 | 0 | 0 | 2
    Asian - South East Asian Heritage | 0 | 5 | 5 | 3 | 13
    White - White/Caucasian/European | 55 | 45 | 39 | 49 | 188

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a >=50% Reduction in Partial-onset Seizure (POS) Frequency From Baseline
Description: The number of participants experiencing a >=50% reduction from Baseline (BL) in POS frequency during the Treatment Phase (TP) (i.e., Titration Phase and Flexible Dose Evaluation [FDE] Phase) was measured. A POS has its onset in a limited area on one side of the brain. POSs may remain limited or may spread to involve both sides of the brain. For both the Baseline Phase and the TP, seizure frequency was calculated as a 28-day rate using the following formula: 28 x {[(number of countable partial seizures in Phase) + (10 x number of days with innumerable seizures in Phase) + (number of occurrences of status epilepticus in Phase)] / number of applicable days in the Phase}, where all days in the Phase are considered applicable (including days with 0 seizures), except for days on which the participant failed to complete the Seizure Diary. >= 50% reduction from BL is calculated as 100 x (28-day partial seizure rate [PSR] for the TP - 28-day PSR for the BL Phase) / 28-day PSR for the BL Phase.
Time Frame: From Baseline through Week 20 (Day 140)/Early Withdrawal
Population: Intent-to-Treat (ITT) Population: all participants in the Safety Population (all participants who took at least one dose of investigational product) who provided at least one post-Baseline efficacy assessment
Measure: Number; unit: participants
Groups:
- Total: All four antiepileptic drug treatment arms combined
Arm/Group | RTG Flexible Dose Plus C/O | RTG Flexible Dose Plus Lamotrigine | RTG Flexible Dose Plus Levetiracetam | RTG Flexible Dose Plus Valproic Acid | Total
Number analyzed (Participants) | 55 | 50 | 44 | 51 | 200
participants | 22 | 16 | 22 | 29 | 89
Statistical Analysis 1: Comparison: RTG Flexible Dose Plus C/O; Test type: Superiority or Other; percentage of participants = 40.0, 95% CI 2-sided [27.1 to 52.9] — The estimated value represents the percentage of participants with a >=50% reduction in partial-onset seizure frequency from Baseline
Statistical Analysis 2: Comparison: RTG Flexible Dose Plus Lamotrigine; Test type: Superiority or Other; percentage of participants = 32.0, 95% CI 2-sided [19.1 to 44.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: RTG Flexible Dose Plus Levetiracetam; Test type: Superiority or Other; percentage of participants = 50.0, 95% CI 2-sided [35.2 to 64.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: RTG Flexible Dose Plus Valproic Acid; Test type: Superiority or Other; percentage of participants = 56.9, 95% CI 2-sided [43.3 to 70.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Total; Test type: Superiority or Other; percentage of participants = 44.5, 95% CI 2-sided [37.6 to 51.4] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Number of Participants With the Indicated Reduction or Increase From Baseline in Partial-onset Seizure Frequency
Description: Participants were assessed for the percent change from Baseline in seizure frequency; changes were categorized as Any Decrease (>0 to 25%, 25 to <50%, 50 to 75%, >75 to 100%) or No Change or Any Increase (>25%, 0 to 25%). A partial-onset seizure is a seizure that has its onset in a limited area on one side of the brain. Partial-onset seizures may remain limited or may spread to involve both sides of the brain.
Time Frame: From Baseline through Week 20 (Day 140)/Early Withdrawal
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | RTG Flexible Dose Plus C/O | RTG Flexible Dose Plus Lamotrigine | RTG Flexible Dose Plus Levetiracetam | RTG Flexible Dose Plus Valproic Acid | Total
Number analyzed (Participants) | 55 | 50 | 44 | 51 | 200
participants
  Any decrease | 43 | 43 | 36 | 44 | 166
  >0 to <25% decrease | 16 | 10 | 6 | 7 | 39
  25 to <50% decrease | 5 | 17 | 8 | 8 | 38
  50 to 75% decrease | 10 | 8 | 14 | 17 | 49
  >75 to 100% decrease | 12 | 8 | 8 | 12 | 40
  No change or any increase | 12 | 7 | 8 | 7 | 34
  >25% increase | 10 | 4 | 5 | 6 | 25
  0 to 25% increase | 2 | 3 | 3 | 1 | 9

3. Secondary Outcome: Number of Participants With a >=25%, >=75%, or 100% Reduction in Partial-onset Seizure Frequency From Baseline
Description: The number of participants experiencing a >=25%, >=75%, and 100% reduction from Baseline in partial-onset seizure frequency during the Treatment Phase (TP) (i.e., Titration Phase and Flexible Dose Evaluation [FDE] Phase) was measured. A partial-onset seizure is a seizure that has its onset in a limited area on one side of the brain. Partial-onset seizures may remain limited or may spread to involve both sides of the brain.
Time Frame: From Baseline through Week 20 (Day 140)/Early Withdrawal
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | RTG Flexible Dose Plus C/O | RTG Flexible Dose Plus Lamotrigine | RTG Flexible Dose Plus Levetiracetam | RTG Flexible Dose Plus Valproic Acid | Total
Number analyzed (Participants) | 55 | 50 | 44 | 51 | 200
participants
  >=25% | 27 | 33 | 30 | 37 | 127
  >=75% | 12 | 8 | 8 | 12 | 40
  100% | 0 | 2 | 1 | 2 | 5

4. Secondary Outcome: Percent Change From Baseline in Partial-onset Seizure Frequency
Description: Percent change from Baseline was calculated as the difference in the partial-onset seizure frequency (Treatment Phase minus the Baseline Phase) divided by the Baseline Phase frequency, multiplied by 100. Negative values indicate reductions from Baseline. A partial-onset seizure is a seizure that has its onset in a limited area on one side of the brain. Partial-onset seizures may remain limited or may spread to involve both sides of the brain.
Time Frame: From Baseline through Week 20 (Day 140)/Early Withdrawal
Population: ITT Population
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | RTG Flexible Dose Plus C/O | RTG Flexible Dose Plus Lamotrigine | RTG Flexible Dose Plus Levetiracetam | RTG Flexible Dose Plus Valproic Acid | Total
Number analyzed (Participants) | 55 | 50 | 44 | 51 | 200
percent change | -24.6 (55.25) | -27.8 (59.97) | -28.7 (80.27) | -27.1 (102.10) | -27.0 (75.68)

5. Secondary Outcome: Functional Status Diary (FSD): Percent Change From Baseline in Epilepsy-related Worry
Description: Participants were asked the following question daily: "How would you rate your epilepsy-related worry over the last 24 hours?" The original possible responses were 0-10, with 0="No worry" and 10="Worst worry imaginable." However, in the summarization, "1" was added to each participant's daily response, changing the possible values to 1-11, so that there would be no possibility of the percent change from Baseline being undefined. Baseline and Treatment Phase averages were calculated for each participant. The denominators for these by-phase averages were the number of non-missing days for each variable and phase. The by-phase averages were used as follows in the calculation of percent change from Baseline for each participant: 100 x Treatment Phase average - Baseline Phase average) / Baseline Phase average. A negative percent change from Baseline indicates a reduction from Baseline.
Time Frame: Baseline through Week 20/Early Withdrawal
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | RTG Flexible Dose Plus C/O | RTG Flexible Dose Plus Lamotrigine | RTG Flexible Dose Plus Levetiracetam | RTG Flexible Dose Plus Valproic Acid | Total
Number analyzed (Participants) | 55 | 50 | 39 | 48 | 192
Percent change | 0.8 (45.60) | -7.5 (29.53) | -9.1 (36.76) | -2.0 (73.16) | -4.1 (49.13)

6. Secondary Outcome: Functional Status Diary (FSD): Percent Change From Baseline in Epilepsy-related Limitation of Ability to do What You Needed to
Description: Participants were asked the following question daily: "How would you rate the extent to which epilepsy limited your ability to do what you needed to do over the last 24 hours?" The original possible responses were 0-10, with 0="Not at all limited" and 10="Unable to do anything I needed to." However, in the summarization, "1" was added to each participant's daily response, changing the possible values to 1-11, so that there would be no possibility of the percent change from Baseline being undefined. Baseline and Treatment Phase averages were calculated for each participant. The denominators for these by-phase averages were the number of non-missing days for each variable and phase. The by-phase averages were used as follows in the calculation of percent change from Baseline for each participant: 100 x Treatment Phase average - Baseline Phase average) / Baseline Phase average. A negative percent change from Baseline indicates a reduction from Baseline.
Time Frame: Baseline through Week 20/Early Withdrawal
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | RTG Flexible Dose Plus C/O | RTG Flexible Dose Plus Lamotrigine | RTG Flexible Dose Plus Levetiracetam | RTG Flexible Dose Plus Valproic Acid | Total
Number analyzed (Participants) | 55 | 50 | 40 | 48 | 193
Percent change | 10.2 (83.80) | -7.7 (25.24) | 2.5 (30.97) | 10.6 (98.84) | 4.1 (69.15)

7. Secondary Outcome: Functional Status Diary (FSD): Percent Change From Baseline in Epilepsy-related Limitation of Ability to do What You Wanted to
Description: Participants were asked the following question daily: "How would you rate the extent to which epilepsy limited your ability to do what you wanted to do over the last 24 hours?" The original possible responses were 0-10, with 0="Not at all limited" and 10="Unable to do anything I wanted to." However, in the summarization, "1" was added to each participant's daily response, changing the possible values to 1-11, so that there would be no possibility of the percent change from Baseline being undefined. Baseline and Treatment Phase averages were calculated for each participant. The denominators for these by-phase averages were the number of non-missing days for each variable and phase. The by-phase averages were used as follows in the calculation of percent change from Baseline for each participant: 100 x Treatment Phase average - Baseline Phase average) / Baseline Phase average. A negative percent change from Baseline indicates a reduction from Baseline.
Time Frame: Baseline through Week 20/Early Withdrawal
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | RTG Flexible Dose Plus C/O | RTG Flexible Dose Plus Lamotrigine | RTG Flexible Dose Plus Levetiracetam | RTG Flexible Dose Plus Valproic Acid | Total
Number analyzed (Participants) | 55 | 50 | 39 | 48 | 192
Percent change | 6.3 (83.07) | -5.0 (25.72) | 3.2 (36.94) | 7.1 (97.31) | 2.9 (68.89)

8. Secondary Outcome: Percent Change From Baseline in Functional Status: Percentage of Days With no Missed Work or School Time
Description: Participants were asked the following question daily: "Did you miss any time from work or school in the last 24 hours due to epilepsy?" Possible responses were Yes, No, and NA=Not Applicable (no planned work or school in the last 24 hours). The variable summarized is the percentage of days with no missed work or school. Baseline and Treatment Phase averages were calculated for each participant. The denominators for these by-phase averages were the number of non-missing days for each variable and phase. The by-phase averages were used as follows in the calculation of percent change from Baseline for each participant: 100 x Treatment Phase average - Baseline Phase average) / Baseline Phase average. A positive percent change from Baseline indicates a reduction from Baseline in missed work or school.
Time Frame: Baseline through Week 20/Early Withdrawal
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | RTG Flexible Dose Plus C/O | RTG Flexible Dose Plus Lamotrigine | RTG Flexible Dose Plus Levetiracetam | RTG Flexible Dose Plus Valproic Acid | Total
Number analyzed (Participants) | 34 | 39 | 31 | 29 | 133
Percent change | 53.5 (295.57) | 4.9 (9.37) | 3.7 (29.33) | 4.5 (11.71) | 17.0 (150.18)

9. Secondary Outcome: Change From Baseline in the Short Form 36 Health Survey, Version 2 (SF-36v2) Domain Scores at Week 20/Early Withdrawal
Description: The SF-36v2 health survey is a self-administered, generic, 36-item questionnaire designed to measure 8 domains of functional health status and well-being: physical functioning, role-physical, bodily pain, general health perceptions, vitality, social functioning, role-emotional, and mental health. Each domain is scored from 0 (poorer health) to 100 (better health). Change from Baseline was calculated as the post-Baseline score minus the Baseline score. Positive changes from Baseline indicate improvement.
Time Frame: Baseline through Week 20/Early Withdrawal
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | RTG Flexible Dose Plus C/O | RTG Flexible Dose Plus Lamotrigine | RTG Flexible Dose Plus Levetiracetam | RTG Flexible Dose Plus Valproic Acid | Total
Number analyzed (Participants) | 53 | 46 | 38 | 46 | 183
Scores on a scale
  Physical Functioning | -0.54 (5.461) | 0.89 (6.665) | -0.70 (4.974) | 0.46 (5.465) | 0.04 (5.689)
  Role-Physical | -1.31 (9.563) | 1.04 (9.366) | 0.31 (10.958) | 1.87 (7.644) | 0.42 (9.390)
  Bodily Pain | 0.92 (10.315) | 0.62 (10.925) | 1.28 (8.571) | 2.81 (11.198) | 1.39 (10.324)
  General Health | -0.35 (7.303) | 2.55 (7.240) | 0.68 (6.342) | 2.45 (7.749) | 1.30 (7.269)
  Vitality | -2.94 (10.657) | 0.52 (9.722) | 0.47 (6.838) | 1.56 (8.318) | -0.23 (9.253)
  Social Functioning | -1.83 (12.022) | 0.58 (11.063) | 1.84 (9.787) | 2.10 (10.107) | 0.53 (10.904)
  Role-Emotional | -1.43 (13.224) | 1.07 (10.991) | 2.19 (9.258) | 4.36 (12.719) | 1.41 (11.915)
  Mental Health | -2.04 (10.510) | 0.72 (9.480) | 2.48 (8.685) | 3.31 (10.636) | 0.94 (10.079)

10. Secondary Outcome: Change From Baseline in the SF-36v2 Physical Component Summary Score at Week 20/Early Withdrawal
Description: The SF-36 v2 Health Survey is a self-administered, generic, 36-item questionnaire designed to measure 8 domains of functional health status and well-being: physical functioning, role-physical, bodily pain, general health perceptions, vitality, social functioning, role-emotional, and mental health. Each domain is scored from 0 (poorer health) to 100 (better health).The physical component summary (PCS) score is a summary score representing overall physical health, which is derived from the 8 domains. As with the domains, PCS scores range from 0 to 100; higher scores represent better health. Change from Baseline was calculated as the post-Baseline score minus the Baseline score. Positive changes from Baseline indicate improvement.
Time Frame: Baseline through Week 20/Early Withdrawal
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | RTG Flexible Dose Plus C/O | RTG Flexible Dose Plus Lamotrigine | RTG Flexible Dose Plus Levetiracetam | RTG Flexible Dose Plus Valproic Acid | Total
Number analyzed (Participants) | 53 | 46 | 38 | 46 | 183
Scores on a scale | 0.17 (5.202) | 1.22 (6.218) | -0.58 (5.648) | 0.82 (4.525) | 0.44 (5.410)

11. Secondary Outcome: Change From Baseline in the SF-36v2 Mental Component Summary Score at Week 20/Early Withdrawal
Description: The SF-36 v2 Health Survey is a self-administered, generic, 36-item questionnaire designed to measure 8 domains of functional health status and well-being: physical functioning, role-physical, bodily pain, general health perceptions, vitality, social functioning, role-emotional, and mental health. Each domain is scored from 0 (poorer health) to 100 (better health).The mental component summary (MCS) score is a summary score representing overall mental health, which is derived from the 8 domains. As with the domains, MCS scores range from 0 to 100; higher scores represent better health. Change from Baseline was calculated as the post-Baseline score minus the Baseline score. Positive changes from Baseline indicate improvement.
Time Frame: Baseline through Week 20/Early Withdrawal
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | RTG Flexible Dose Plus C/O | RTG Flexible Dose Plus Lamotrigine | RTG Flexible Dose Plus Levetiracetam | RTG Flexible Dose Plus Valproic Acid | Total
Number analyzed (Participants) | 53 | 46 | 38 | 46 | 183
Scores on a scale | -2.59 (12.359) | 0.66 (10.149) | 2.75 (8.851) | 3.79 (10.206) | 0.94 (10.825)

12. Secondary Outcome: Number of Participants With the Indicated Response for the Epilepsy-related Worry Component of the Patient Global Impression of Change (PGI-C) Score
Description: The PGI-C questionnaire was to be completed by the participant. Participants were asked the following question: Compared to before you started this study, how would you rate your current epilepsy-related worry: Much better, Moderately better, A little better, Unchanged, A little worse, Moderately worse, Much worse?
Time Frame: Baseline through Week 20/Early Withdrawal
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: participants
Arm/Group | RTG Flexible Dose Plus C/O | RTG Flexible Dose Plus Lamotrigine | RTG Flexible Dose Plus Levetiracetam | RTG Flexible Dose Plus Valproic Acid | Total
Number analyzed (Participants) | 53 | 46 | 40 | 46 | 185
participants
  Much better | 7 | 9 | 4 | 11 | 31
  Moderately better | 11 | 16 | 15 | 16 | 58
  A little better | 13 | 6 | 4 | 11 | 34
  Unchanged | 16 | 11 | 13 | 6 | 46
  A little worse | 5 | 2 | 4 | 0 | 11
  Moderately worse | 0 | 1 | 0 | 0 | 1
  Much worse | 1 | 1 | 0 | 2 | 4

13. Secondary Outcome: Change From Baseline in the PGI-C Score: Epilepsy-related Worry
Description: The PGI-C questionnaire was to be completed by the participant. Participants were asked the following question: Compared to before you started this study, how would you rate your current epilepsy-related worry: Much better, Moderately better, A little better, Unchanged, A little worse, Moderately worse, Much worse? Rating scores are integers from 1 to 7, with 1=Much better and 7=Much worse.
Time Frame: Baseline through Week 20/Early Withdrawal
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | RTG Flexible Dose Plus C/O | RTG Flexible Dose Plus Lamotrigine | RTG Flexible Dose Plus Levetiracetam | RTG Flexible Dose Plus Valproic Acid | Total
Number analyzed (Participants) | 53 | 46 | 40 | 46 | 185
Scores on a scale | 3.1 (1.32) | 2.7 (1.44) | 3.0 (1.24) | 2.5 (1.38) | 2.8 (1.36)

14. Secondary Outcome: Number of Participants With the Indicated Response for the Current Ability to do the Things You Need to do Component of the PGI-C Score
Description: The PGI-C questionnaire was to be completed by the participant. Participants were asked the following question: Compared to before you started this study, how would you rate your current ability to do the things you need to do: Much better, Moderately better, A little better, Unchanged, A little worse, Moderately worse, Much worse?
Time Frame: Baseline through Week 20/Early Withdrawal
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: participants
Arm/Group | RTG Flexible Dose Plus C/O | RTG Flexible Dose Plus Lamotrigine | RTG Flexible Dose Plus Levetiracetam | RTG Flexible Dose Plus Valproic Acid | Total
Number analyzed (Participants) | 53 | 46 | 40 | 46 | 185
participants
  Much better | 5 | 9 | 6 | 10 | 30
  Moderately better | 13 | 11 | 9 | 14 | 47
  A little better | 10 | 6 | 6 | 9 | 31
  Unchanged | 19 | 17 | 17 | 11 | 64
  A little worse | 2 | 3 | 1 | 1 | 7
  Moderately worse | 2 | 0 | 0 | 0 | 2
  Much worse | 2 | 0 | 1 | 1 | 4

15. Secondary Outcome: Change From Baseline in the PGI-C Score: Current Ability to do the Things You Need to do
Description: The PGI-C questionnaire was to be completed by the participant. Participants were asked the following question: Compared to before you started this study, how would you rate your current ability to do the things you need to do: Much better, Moderately better, A little better, Unchanged, A little worse, Moderately worse, Much worse? Rating scores are integers from 1 to 7, with 1=Much better and 7=Much worse.
Time Frame: Baseline through Week 20/Early Withdrawal
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | RTG Flexible Dose Plus C/O | RTG Flexible Dose Plus Lamotrigine | RTG Flexible Dose Plus Levetiracetam | RTG Flexible Dose Plus Valproic Acid | Total
Number analyzed (Participants) | 53 | 46 | 40 | 46 | 185
Scores on a scale | 3.3 (1.43) | 2.9 (1.29) | 3.1 (1.34) | 2.6 (1.32) | 3.0 (1.36)

16. Secondary Outcome: Number of Participants With the Indicated Response for the Current Ability to do the Things You Want to do Component of the PGI-C Score
Description: The PGI-C questionnaire was to be completed by the participant. Participants were asked the following question: Compared to before you started this study, how would you rate your current ability to do the things you want to do: Much better, Moderately better, A little better, Unchanged, A little worse, Moderately worse, Much worse.
Time Frame: Baseline through Week 20/Early Withdrawal
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: participants
Arm/Group | RTG Flexible Dose Plus C/O | RTG Flexible Dose Plus Lamotrigine | RTG Flexible Dose Plus Levetiracetam | RTG Flexible Dose Plus Valproic Acid | Total
Number analyzed (Participants) | 53 | 46 | 40 | 46 | 185
participants
  Much better | 2 | 8 | 4 | 11 | 25
  Moderately better | 13 | 13 | 12 | 16 | 54
  A little better | 11 | 4 | 6 | 9 | 30
  Unchanged | 20 | 20 | 17 | 8 | 65
  A little worse | 3 | 1 | 1 | 1 | 6
  Moderately worse | 3 | 0 | 0 | 0 | 3
  Much worse | 1 | 0 | 0 | 1 | 2

17. Secondary Outcome: Change From Baseline in the PGI-C Score: Current Ability to do the Things You Want to do
Description: The PGI-C questionnaire was to be completed by the participant. Participants were asked the following question: Compared to before you started this study, how would you rate your current ability to do the things you want to do: Much better, Moderately better, A little better, Unchanged, A little worse, Moderately worse, Much worse? Rating scores are integers from 1 to 7, with 1=Much better and 7=Much worse.
Time Frame: Baseline through Week 20/Early Withdrawal
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | RTG Flexible Dose Plus C/O | RTG Flexible Dose Plus Lamotrigine | RTG Flexible Dose Plus Levetiracetam | RTG Flexible Dose Plus Valproic Acid | Total
Number analyzed (Participants) | 53 | 46 | 40 | 46 | 185
Scores on a scale | 3.4 (1.29) | 2.8 (1.23) | 3.0 (1.12) | 2.5 (1.30) | 2.9 (1.28)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of study medication through the end of the Follow-up Phase (up to Week 33). SAEs considered to be related to study participation were also to be collected prior to treatment.
Description: SAEs and non-serious AEs were collected in members of the Safety Population, comprised of all participants who took at least one dose of investigational product.
Arm/Group | RTG Flexible Dose Plus C/O | RTG Flexible Dose Plus Lamotrigine | RTG Flexible Dose Plus Levetiracetam | RTG Flexible Dose Plus Valproic Acid
Serious Adverse Events (participants affected / at risk) | 0/56 | 4/51 | 4/44 | 1/52
Other Adverse Events (participants affected / at risk) | 39/56 | 33/51 | 23/44 | 31/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RTG Flexible Dose Plus C/O (N=56) | RTG Flexible Dose Plus Lamotrigine (N=51) | RTG Flexible Dose Plus Levetiracetam (N=44) | RTG Flexible Dose Plus Valproic Acid (N=52)
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 1 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Partial seizures (Nervous system disorders) | 0 | 1 | 0 | 0
Partial seizures with secondary generalization (Nervous system disorders) | 0 | 1 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 1 | 0
Vestibular disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RTG Flexible Dose Plus C/O (N=56) | RTG Flexible Dose Plus Lamotrigine (N=51) | RTG Flexible Dose Plus Levetiracetam (N=44) | RTG Flexible Dose Plus Valproic Acid (N=52)
Dizziness (Nervous system disorders) | 15 | 15 | 14 | 9
Somnolence (Nervous system disorders) | 11 | 8 | 7 | 17
Vertigo (Ear and labyrinth disorders) | 5 | 7 | 3 | 4
Fatigue (General disorders) | 6 | 5 | 5 | 1
Asthenia (General disorders) | 1 | 2 | 5 | 4
Disturbance in attention (Nervous system disorders) | 3 | 3 | 0 | 3
Headache (Nervous system disorders) | 1 | 4 | 2 | 2
Memory impairment (Nervous system disorders) | 4 | 1 | 1 | 2
Speech disorder (Nervous system disorders) | 2 | 4 | 2 | 0
Confusional state (Psychiatric disorders) | 3 | 0 | 3 | 1
Nausea (Gastrointestinal disorders) | 2 | 4 | 1 | 0
Convulsion (Nervous system disorders) | 1 | 1 | 1 | 3
Diplopia (Eye disorders) | 3 | 0 | 1 | 0
Ataxia (Nervous system disorders) | 3 | 0 | 0 | 0
Strangury (Renal and urinary disorders) | 3 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.